CLINICAL TRIAL: NCT02340585
Title: Safety and Effectiveness of the Treatment of Wide Neck, Intracranial, Saccular Aneurysms With the Next Generation Neuroform Stent System
Brief Title: Neuroform Atlas Stent System Study
Acronym: ATLAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Neurovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATLAS
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Results first posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Intracranial Aneurysm
Keywords: Next Generation Neuroform Stent System; Wide Neck, Intracranial, Saccular Aneurysms; Cerebral Aneurysms
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Next Generation Neuroform Stent System (Experimental): The Next Generation Stent System is a self-expanding, open cell, nitinol stent designed to provide support of the coil mass within the aneurysm and minimize stent deflection.
  Interventions: Device: Next Generation Neuroform Stent System

INTERVENTIONS:
Device: Next Generation Neuroform Stent System — The Next Generation Neuroform Stent System is pre-loaded on a stent delivery wire and protected by a transfer sheath. An accessory pouch containing an optional stabilizer may be attached to the proximal end of the stent delivery wire to facilitate handling and stabilization.

SUMMARY:
The primary objective of this study is to demonstrate effectiveness and safety of the Neuroform Atlas Stent System for use with bare metal embolic coils.

DETAILED DESCRIPTION:
The study is a prospective, multicenter, open-label, single arm trial designed to demonstrate the potential treatment of wide neck, intracranial, saccular aneurysms with the Next Generation Neuroform Stent System with any approved embolic coils currently on the market. The study will evaluate the percent occlusion of the treated target lesion on angiography in the absence of retreatment, or parent artery stenosis at the target location at 12 months. Subjects with documented wide neck, intracranial, saccular aneurysms arising from a parent artery may potentially benefit from stent assisted coiling, provided they meet the other eligibility criteria.

Data collected through the 12-month follow-up visit are intended to support Premarket Approval (PMA) application to the Food and Drug Administration (FDA). Long-term follow-up data collected through 3 years postoperative are intended to support post-approval study (PAS) requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 18 and 80 years of age
2. Documented wide neck (neck ≥ 4 mm or a dome-to-neck ratio of < 2), intracranial, saccular aneurysm arising from a parent vessel with a diameter of ≥ 2mm and ≤ 4.5 mm, which will be treated with bare metal coils
3. Subject or legal representative is willing and able to provide informed consent
4. Subject is willing and able to comply with protocol follow-up requirements

Exclusion Criteria:

1. Known multiple untreated cerebral aneurysms, other than non-target blister aneurysm, infundibulum, or aneurysm measuring <3mm for each of three dimensions assessed (height, width, and depth) that will not require treatment during the study period
2. Target lesion is a blister aneurysm, infundibulum, or aneurysm measuring <3mm for each of three dimensions assessed (height, width, and depth)
3. Target aneurysm that will require an Investigator to intentionally leave a neck remnant in order to preserve blood flow in a bifurcation or branch
4. Coiling or stenting of a non-target intracranial aneurysm within 30 days prior to study treatment
5. Target aneurysm is in the anterior circulation proximal to the superior hypophyseal ICA
6. Acute target aneurysm rupture less than 14 days prior to study treatment
7. Hunt and Hess score ≥ 3 or a premorbid mRS score ≥4
8. An admission platelet count of <50,000, any known coagulopathy, or an International Normalized Ratio (INR)>3.0 without oral anticoagulation therapy
9. A known absolute contraindication to angiography
10. Evidence of active cancer, terminal illness or any condition which, in the opinion of the treating physician, would/could prevent subject from completing the study (e.g., a high risk of embolic stroke, atrial fibrillation, co-morbidities, psychiatric disorders, substance abuse, major surgery ≤ 30 days pre-procedure, etc.)
11. Known absolute contraindication to the use of required study medications or agents (e.g., heparin, aspirin, clopidogrel, and radiographic contrast agents, etc.)
12. Female subject who is pregnant or intends to become pregnant during the study
13. Moya-Moya disease, arteriovenous malformation(s), arteriovenous fistula(e), intracranial tumor(s), or intracranial hematoma(s) (unrelated to target aneurysm)
14. Significant atherosclerotic stenosis, significant vessel tortuosity, vasospasm refractory to medication, unfavorable aneurysm morphology or vessel anatomy, or some other condition(s) that, in the opinion of the treating physician, would/could prevent or interfere with access to the target aneurysm and/or successful deployment of the Neuroform Atlas™ Stent
15. Previous treatment (e.g., surgery, stenting) in the parent artery that, in the opinion of the treating physician, would/could prevent or interfere with successful use of the Neuroform Atlas™ Stent System and/or successful adjunctive deployment of embolic coils
16. Previous stent-assisted coiling of the target aneurysm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2015-06-18 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Osama Zaidat, MD, Principal Investigator — Mercy Health - St. Vincent Medical Center; Brian Jankowitz, MD, Principal Investigator — Cooper University Health Center
Locations (25):
- United States (25):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Vascular Neurology of Southern California, Thousand Oaks, California
  - Radiology Imaging Associates, Englewood, Colorado
  - Christiana Care Health Services, Newark, Delaware
  - Lyerly Neurosurgery, Jacksonville, Florida
  - WellStar Kennestone Hospital, Marietta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Kentucky Research Foundation, Lexington, Kentucky
  - The Johns Hopkins University, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - SSM Health DePaul Hospital, Bridgeton, Missouri
  - SUNY University at Buffalo Neurosurgery/Gates Vascular Institute, Buffalo, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Mercy Health - St. Vincent Medical Center, Toledo, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Methodist Healthcare - Memphis Hospitals, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Hanel RA, Cortez GM, Jankowitz BT, Sauvageau E, Aghaebrahim A, Lin E, Jadhav AP, Gross B, Khaldi A, Gupta R, Frei D, Loy D, Price LL, Hetts SW, Zaidat OO; ATLAS Investigators. Anterior circulation location-specific results for stent-assisted coiling - carotid versus distal aneurysms: 1-year outcomes from the Neuroform Atlas Stent Pivotal Trial. J Neurointerv Surg. 2024 Oct 14;16(11):1125-1130. doi: 10.1136/jnis-2023-020591. PMID 37940387
- [Derived] Jankowitz BT, Jadhav AP, Gross B, Jovin TG, Alhajeri AA, Fraser JF, Hanel RA, Sauvageau E, Aghaebrahim A, Frei D, Bellon R, Loy D, Puri AS, Malek AM, Thomas A, Toth G, Lopes DK, Crowley RW, Arthur AS, Reavey-Cantwell J, Lin E, Siddiqui AH, Alexander MJ, Khaldi A, Colby GP, Caplan JM, Satti SR, Turk AS, Spiotta AM, Klucznik R, Hallam DK, Kung D, Froehler MT, Callison RC, Kan P, Hetts SW, Zaidat OO. Pivotal trial of the Neuroform Atlas stent for treatment of posterior circulation aneurysms: one-year outcomes. J Neurointerv Surg. 2022 Feb;14(2):143-148. doi: 10.1136/neurintsurg-2020-017115. Epub 2021 Mar 15. PMID 33722961
- [Derived] Zaidat OO, Hanel RA, Sauvageau EA, Aghaebrahim A, Lin E, Jadhav AP, Jovin TG, Khaldi A, Gupta RG, Johnson A, Frei D, Loy D, Malek A, Toth G, Siddiqui A, Reavey-Cantwell J, Thomas A, Hetts SW, Jankowitz BT; ATLAS Investigators. Pivotal Trial of the Neuroform Atlas Stent for Treatment of Anterior Circulation Aneurysms: One-Year Outcomes. Stroke. 2020 Jul;51(7):2087-2094. doi: 10.1161/STROKEAHA.119.028418. Epub 2020 Jun 17. PMID 32568654

RESULTS

PARTICIPANT FLOW:
Period: Anterior Cohort
Arm/Group | Next Generation Neuroform Stent System
Started | 182
Completed | 182
Not Completed | 0
Period: Posterior Cohort
Arm/Group | Next Generation Neuroform Stent System
Started | 116
Completed | 116
Not Completed | 0
Period: Post-approval Study (PAS)
Arm/Group | Next Generation Neuroform Stent System
Started | 298
Completed | 298
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Next Generation Neuroform Stent System
Number analyzed (Participants) | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 227
  Male | 71
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 253
  black | 34
  Asian | 5
  Native Hawaiian or other Pacific Islander | 1
  American Indian or Alaskan Native | 1
  Other | 4

OUTCOME MEASURES:

1. Primary Outcome: Stroke or Death
Description: Any major ipsilateral stroke or neurological death
Time Frame: within 12 months of the index procedure
Measure: Count of Participants; unit: Participants
Groups:
- Neuroform Atlas Stent System (Anterior): Neuroform Atlas Stent System (Anterior)
- Neuroform Atlas Stent System (Posterior): Neuroform Atlas Stent System (Posterior)
Arm/Group | Neuroform Atlas Stent System (Anterior) | Neuroform Atlas Stent System (Posterior)
Number analyzed (Participants) | 182 | 116
Participants | 8 | 5

2. Primary Outcome: Aneurysm Occlusion of the Treated Target Lesion on 12 Month Angiography
Description: Complete aneurysm occlusion (100% occlusion - Raymond Class 1) of the treated target lesion on 12 month angiography, in the absence of retreatment, or parent artery stenosis (> 50%) at the target location.
Time Frame: 12 month post index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Neuroform Atlas Stent System (Anterior) | Neuroform Atlas Stent System (Posterior)
Number analyzed (Participants) | 153 | 95
Participants | 135 | 81

3. Secondary Outcome: The Percent of Subjects Experiencing One or More Serious Adverse Events (SAEs) Through 12 Months
Description: The percent of subjects experiencing one or more serious adverse events (SAEs) through 12 months including
  * New or worsening major ipsilateral stroke as measured by the National Institute of Health Stroke Scale (NIHSS)
  * Device-related SAEs
  * Subarachnoid hemorrhage (SAH)
  * Aneurysm rupture
Time Frame: within 12 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Neuroform Atlas Stent System (Anterior) | Neuroform Atlas Stent System (Posterior)
Number analyzed (Participants) | 182 | 116
Participants | 20 | 19

ADVERSE EVENTS:
Time Frame: 12 months
Description: Serious AE, Non-serious AE, All AE
Arm/Group | Next Generation Neuroform Stent System
All-Cause Mortality (participants affected / at risk) | 2/298
Serious Adverse Events (participants affected / at risk) | 90/298
Other Adverse Events (participants affected / at risk) | 212/298
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Next Generation Neuroform Stent System (N=298)
Cerebral artery embolism (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 11 (11)
Subarachnoid haemorrhage (Nervous system disorders) | 5 (5)
Transient ischaemic attack (Nervous system disorders) | 7 (9)
Myelodysplastic Syndrome (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Chest pain (General disorders) | 5 (5)
Myocardial infarction (Cardiac disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Blurred vision (Eye disorders) | 2 (2)
Diplopia (Eye disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis ischemic (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1)
Diarrheic (Gastrointestinal disorders) | 1 (1)
Diverticulitis intestinal hemmorhagic (Gastrointestinal disorders) | 1 (1)
Gastrointestinal hemmorhage (Gastrointestinal disorders) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Application site hematoma (General disorders) | 3 (3)
Hematemesis (Gastrointestinal disorders) | 1 (1)
Human anaplasmosis (Infections and infestations) | 1 (1)
Enterocolitis viral (Infections and infestations) | 1 (1)
Groin infection (Infections and infestations) | 1 (1)
Pelvic abcess (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2)
Post-procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Subdural hematoma (Injury, poisoning and procedural complications) | 2 (2)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1)
vessel perforation (Injury, poisoning and procedural complications) | 1 (1)
Inappropriate antidiurectic hormone secretion (Metabolism and nutrition disorders) | 1 (1)
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle hemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Neck pain (Metabolism and nutrition disorders) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1)
Convulsion or seizure (Nervous system disorders) | 4 (4)
Migraine or status migrainosis (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (2)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Parathesia (Nervous system disorders) | 1 (1)
Vertebral artery dissection (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1)
Ruptured cerebral aneurysm (Nervous system disorders) | 2 (2)
Speech disorder (Nervous system disorders) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Acute prerenal failure (Renal and urinary disorders) | 1 (1)
Nephrogenic anemia (Renal and urinary disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Carotid artery stent insertion (Surgical and medical procedures) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Angioplasty (Surgical and medical procedures) | 1 (1)
Intracerebral aneurysm operation (Surgical and medical procedures) | 18 (20)
Colostomy (Surgical and medical procedures) | 1 (1)
Peripheral artery stent insertion (Surgical and medical procedures) | 1 (1)
Spinal operation (Surgical and medical procedures) | 1 (1)
Peripheral ischemia (Vascular disorders) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 1 (1)
Carotid artery stenosis (Vascular disorders) | 1 (1)
Retroperitoneal hemorrhage (Vascular disorders) | 2 (2)
Thrombosis in device (Vascular disorders) | 3 (3)
Arteriosclerosis (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Next Generation Neuroform Stent System (N=298)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Increased tendency to bruise (Blood and lymphatic system disorders) | 7 (7)
Arrhythmia, tachycardia, afib or bradycardia (Cardiac disorders) | 7 (7)
Ear pain (Ear and labyrinth disorders) | 3 (3)
Photophobia (Eye disorders) | 6 (6)
Blurred vision, diplopia, vision impairment or reduced acuity (Eye disorders) | 15 (15)
Vitreous floaters (Eye disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 5 (5)
Abdominal pain or discomfort (Gastrointestinal disorders) | 8 (8)
Nausea or vomiting (Gastrointestinal disorders) | 16 (18)
Application site injury (General disorders) | 19 (19) — Administration site pain, swelling, secretion, hematoma or hemmorhage
Fatigue (General disorders) | 5 (5)
Chest pain (General disorders) | 3 (3)
Asthenia (General disorders) | 3 (3)
Any pain (General disorders) | 7 (8) — chest, facial, application site, general
Infection (Infections and infestations) | 37 (47)
Urinary tract infection (Infections and infestations) | 18 (18)
Respiratory tract infection (Infections and infestations) | 7 (8)
Pneumonia (Infections and infestations) | 3 (3)
Fall (Musculoskeletal and connective tissue disorders) | 7 (8)
Hypokalemia (Metabolism and nutrition disorders) | 8 (9)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Neck pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Other musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 (13) — arthalgia, groin pain, musculoskeletal pain, pain in extremity
Cerebral vasoconstriction (Nervous system disorders) | 26 (27)
Dizziness (Nervous system disorders) | 17 (17)
Convulsion (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 72 (85)
Vertebral artery dissection (Nervous system disorders) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 10 (14)
Transient ischemic attack (Nervous system disorders) | 3 (3)
Hemiparesis (Nervous system disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 6 (6)
Hypertension (Vascular disorders) | 4 (4)
Hypotension (Vascular disorders) | 6 (7)
Contusion (Vascular disorders) | 3 (3)
Thrombosis in device (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/85/NCT02340585/Prot_SAP_000.pdf